CLINICAL TRIAL: NCT02951273
Title: Cerebral Blood Flow During Propofol Anaesthesia
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Niels Damkjær Olesen, MD, Rigshospitalet, Denmark
Other Study IDs: H-16036250
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Gastrointestinal Neoplasms
Keywords: abdominal surgery; blood pressure; cardiac output; cerebral blood flow; cerebral oxygenation; CO2 reactivity; duplex ultrasound; general anaesthesia; mesenteric traction syndrome; near-infrared spectroscopy; upper gastrointestinal cancer surgery
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study of cerebral blood flow: Patients undergoing oesophageal- or ventricular resection (n=30)
  Interventions: Other: Study of cerebral blood flow

INTERVENTIONS:
Other: Study of cerebral blood flow — Measurements are conducted from before induction of anaesthesia and until 2 hours after the start of surgery and include internal carotid artery blood flow, mean arterial pressure, heart rate, stroke volume, cardiac output, total peripheral resistance, forehead skin blood flow and haemoglobin concentrations, depth of anaesthesia, and frontal lobe, skin, and muscle oxygenation. Further measurements are conducted during hyperventilation before induction of anaesthesia and during hypo-, normo- and hypercapnia during anaesthesia.
  Blood samples are obtained from the arterial line for evaluation of the arterial CO2 tension and markers of mesenteric traction syndrome. Total volume of blood sampled is less than 75 ml.

SUMMARY:
General anaesthesia often reduces blood pressure whereby blood flow to the brain and other vital organs may become insufficient. Thus, medicine is often administered during anaesthesia to maintain blood pressure. However, it is unclear at what level blood pressure should be aimed at during anaesthesia.

Several factors may affect blood flow to the brain during anaesthesia. During surgery on the internal organs, a hormone may be released that dilates blood vessels and causes a so-called mesenteric traction syndrome characterised by a decrease in blood pressure and flushing. This reaction lasts for approximately thirty minutes and is observed in about half of the patients who undergo surgery on the stomach and intestines. It is unknown whether a mesenteric traction syndrome affects blood flow to the brain. Ventilation is also of importance for blood flow to the brain. Thus, blood flow to the brain is reduced by hyperventilation and increases if breathing is slower. It is unclear whether the relation between blood flow to the brain and ventilation is affected during anaesthesia.

This study will evaluate how blood flow to the brain is affected by anaesthesia and standard treatment of a possible reduction in blood pressure. Further, the study will assess whether blood flow to the brain is affected by development of a mesenteric traction syndrome. Lastly, the project will evaluate blood flow to the brain during short-term changes in the patient's ventilation by adjustments on the ventilator.

Thirty patients planned for major abdominal surgery will be included in the project. The study will take place from the patient's arrival at the operation room and until two hours after the start of surgery. Placement of catheters and anaesthesia are according to standard care. Blood flow to the brain will be evaluated using ultrasound. Oxygenation of the brain, skin and muscle will be evaluated by probes that emit light. Depth of anaesthesia is assessed by recording the electrical activity of the brain. Blood pressure is measured by a catheter placed in an artery at the wrist and blood samples will be drawn from the catheter.

DETAILED DESCRIPTION:
Background General anaesthesia reduces blood pressure, but cerebral autoregulation is considered to maintain its blood flow if mean arterial pressure (MAP) is between 60-150 mmHg. Thus, vasoactive medication is administered to treat anaesthesia-induced hypotension if MAP decreases to below approximately 60 mmHg. In young healthy adults, propofol anaesthesia, with limited reduction in blood pressure, decreases cerebral blood flow by approximately 50% by a decrease in neuronal activity. However, it is unknown whether the anaesthesia-induced reduction in cerebral blood flow is affected by a marked decrease in MAP and whether propofol anaesthesia affects the lower level of cerebral autoregulation.

If central blood volume is maintained, cerebral oxygenation may be unaffected by a decrease in MAP to ~40 mmHg whereas a reduction in central blood volume and cardiac output (CO) during orthostasis or bleeding, reduces cerebral oxygenation when MAP is lower than approximately 80 mmHg. Thus, CO may affect cerebral blood flow and the ability to increase CO is likely of importance for maintaining a sufficient cerebral blood flow.

During anaesthesia, cerebral blood flow and MAP may be affected by various factors including release of vasoactive substances. Manipulation of the abdominal organs may induce a so-called mesenteric traction syndrome (MTS) encompassing a triad of flushing, hypotension, and tachycardia in about half of the patients who undergo major abdominal surgery. MTS typically develops 15-20 min after the start of surgery and the haemodynamic manifestations, that appear to be mediated by prostaglandin I2, last for approximately 30 min. The effect of MTS on cerebral blood flow is unknown. Prostaglandin I2 dilates cerebral arteries in vitro but does not affect cerebral blood flow when administered to healthy subjects. In a previous study we found that MTS increases near-infrared spectroscopy determined frontal lobe oxygenation possibly due to an increase in extracranial circulation while there was no effect on middle cerebral artery mean flow velocity as an index of changes in cerebral blood flow.

Propofol anaesthesia appears not to affect the CO2 reactivity of the middle cerebral artery as determined by transcranial Doppler ultrasonography, but the CO2 reactivity of the internal carotid artery during propofol anaesthesia is unknown.

Objective The purpose of this study is to evaluate how internal carotid artery blood flow is affected by propofol anaesthesia and related hypotension, and by administration of phenylephrine as standard care to treat anaesthesia-induced hypotension. Further, the study will assess whether internal carotid artery blood flow is affected by development of MTS and whether propofol anaesthesia affects the CO2 reactivity of the internal carotid artery.

Hypotheses

1. Propofol anaesthesia and related anaesthesia-induced hypotension (MAP < 65 mmHg) reduces internal carotid artery blood flow
2. Treatment of anaesthesia-induced hypotension by administration of phenylephrine increases internal carotid artery blood flow
3. Development of MTS increases near-infrared spectroscopy determined frontal lobe oxygenation due to an increase in forehead skin blood flow and oxygenation with no effect on internal carotid artery blood flow
4. Propofol anaesthesia lowers the CO2 reactivity of the internal carotid artery

Methods The study will include thirty patients undergoing oesophageal- or ventricular resection. The study lasts from when the patient arrives to the operating room and until two hours after the start of surgery. As part of standard care all patients will be instrumented with arterial and central venous catheters. Anaesthesia will be induced by propofol and maintained by propofol and remifentanil combined with epidural anaesthesia. Development of MTS is defined by flushing within the first 60 min of surgery. Measurements include unilateral internal carotid artery blood flow evaluated by duplex ultrasound, MAP and heart rate as recorded by a transducer connected to the arterial line, central haemodynamics (stroke volume, CO, and total peripheral resistance) evaluated by pulse contour analysis of the arterial pressure curve, frontal lobe and muscle oxygenation as determined by near-infrared spectroscopy, forehead skin blood flow, haemoglobin concentrations, and oxygenation assessed by laser Doppler flowmetry, and depth of anaesthesia determined by Bispectral Index. At each time point 2 measurements of internal carotid artery blood flow are collected and the mean is taken. Arterial blood will be drawn for analysis of the arterial CO2 tension (PaCO2).

During the study PaCO2 will be maintained at the value before induction of anaesthesia by ventilator adjustments. Internal carotid artery CO2 reactivity before induction of anaesthesia will be determined by evaluations of blood flow and PaCO2 during normoventilation and during hyperventilation to reduce PaCO2 by 1.5 kPa as guided by end-tidal CO2 tension (PetCO2) and measurements will be conducted when PetCO2 has been stable for 5 min. The CO2 reactivity during anaesthesia will be determined by evaluations of internal carotid artery blood flow and PaCO2 at a PaCO2 at the value before induction of anaesthesia and 1.5 kPa above and below that value as guided by PetCO2 and measurements will be conducted when PetCO2 has been stable for 5 min. The CO2 reactivity before and during anaesthesia is calculated as the percentage change in internal carotid artery blood flow per kPa change in PaCO2. Analysis of internal carotid blood flow will be after correction for CO2 reactivity.

Blood samples for analysis of markers of MTS (6-keto-prostaglandin-F1, pro-ANP, ACTH, cortisone, IL-1, IL-6, and TNF-α) will be drawn before induction of anaesthesia and 20 and 60 min after the start of surgery. Total amount of blood samples will be no more than 75 ml. Patients will be excluded if the planned surgery is cancelled and excluded patients will be replaced.

Measurements will be conducted and arterial blood drawn at the following time points:

* Before induction of anaesthesia during normoventilation and hyperventilation
* After induction of anaesthesia
* During anaesthesia-induced hypotension (MAP < 65 mmHg)
* After treatment of anaesthesia-induced hypotension by administration of phenylephrine
* 5 min before and after incision and 0, 20, 40 and 70 min after development of MTS and 20, 40, 60 and 90 min after the start of surgery in patients who did not develop MTS
* During normo-, hyper-, and hypocapnia during anaesthesia in random order

Statistics Trial size: The minimal clinically important difference in internal carotid artery blood flow by treatment of anaesthesia-induced hypotension is considered to be 10%, corresponding to approximately 24 ml/min, and twenty-seven patients were considered required assuming a 42 ml/min SD with a 5% significance level and a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for major abdominal surgery that require placement of an arterial line and central venous catheter, including oesophageal- or ventricular resection
* Age ≥ 18 years.

Exclusion Criteria:

* No informed consent
* Robotic assisted procedures
* Treatment with anti-inflammatory medication, including NSAID and corticosteroids
* Atherosclerosis of the internal carotid artery that obstructs ≥ 30% of the vessel lumen
* Neurologic disease considered to affect cerebral blood flow, including dementia, epilepsy, and apoplexy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients planned for oesophageal- or ventricular resection at Department of Anaesthesia, Rigshospitalet, Copenhagen, Denmark
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niels H. Secher, MD, D.M.Sc., Study Director — Department of Anaesthesia, Rigshospitalet 2043, DK-2100 Copenhagen Ø, Denmark; Niels D. Olesen, MD, Principal Investigator — Department of Anaesthesia, Rigshospitalet 2043, DK-2100 Copenhagen Ø, Denmark
Locations (1):
- Department of Anaesthesia, Rigshospitalet 2043, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fujimoto Y, Nomura Y, Hirakawa K, Hotta A, Nakamoto A, Yoshikawa N, Ohira N, Tatekawa S. Flurbiprofen axetil provides a prophylactic benefit against mesenteric traction syndrome associated with remifentanil infusion during laparotomy. J Anesth. 2012 Aug;26(4):490-5. doi: 10.1007/s00540-012-1368-8. Epub 2012 Mar 2. PMID 22382665
- [Background] Jorgensen LG, Perko M, Perko G, Secher NH. Middle cerebral artery velocity during head-up tilt induced hypovolaemic shock in humans. Clin Physiol. 1993 Jul;13(4):323-36. doi: 10.1111/j.1475-097x.1993.tb00333.x. PMID 8370233
- [Background] Kaisti KK, Metsahonkala L, Teras M, Oikonen V, Aalto S, Jaaskelainen S, Hinkka S, Scheinin H. Effects of surgical levels of propofol and sevoflurane anesthesia on cerebral blood flow in healthy subjects studied with positron emission tomography. Anesthesiology. 2002 Jun;96(6):1358-70. doi: 10.1097/00000542-200206000-00015. PMID 12170048
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, Hert SD, Ford I, Gonzalez-Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luscher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Sousa-Uva M, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur Heart J. 2014 Sep 14;35(35):2383-431. doi: 10.1093/eurheartj/ehu282. Epub 2014 Aug 1. No abstract available. PMID 25086026
- [Background] LASSEN NA. Cerebral blood flow and oxygen consumption in man. Physiol Rev. 1959 Apr;39(2):183-238. doi: 10.1152/physrev.1959.39.2.183. No abstract available. PMID 13645234
- [Background] Matta BF, Lam AM, Strebel S, Mayberg TS. Cerebral pressure autoregulation and carbon dioxide reactivity during propofol-induced EEG suppression. Br J Anaesth. 1995 Feb;74(2):159-63. doi: 10.1093/bja/74.2.159. PMID 7696064
- [Background] Meng L, Hou W, Chui J, Han R, Gelb AW. Cardiac Output and Cerebral Blood Flow: The Integrated Regulation of Brain Perfusion in Adult Humans. Anesthesiology. 2015 Nov;123(5):1198-208. doi: 10.1097/ALN.0000000000000872. PMID 26402848
- [Background] Nissen P, van Lieshout JJ, Nielsen HB, Secher NH. Frontal lobe oxygenation is maintained during hypotension following propofol-fentanyl anesthesia. AANA J. 2009 Aug;77(4):271-6. PMID 19731845
- [Background] Ogoh S, Sato K, Okazaki K, Miyamoto T, Secher F, Sorensen H, Rasmussen P, Secher NH. A decrease in spatially resolved near-infrared spectroscopy-determined frontal lobe tissue oxygenation by phenylephrine reflects reduced skin blood flow. Anesth Analg. 2014 Apr;118(4):823-9. doi: 10.1213/ANE.0000000000000145. PMID 24651237
- [Background] Takada M, Taruishi C, Sudani T, Suzuki A, Iida H. Intravenous flurbiprofen axetil can stabilize the hemodynamic instability due to mesenteric traction syndrome--evaluation with continuous measurement of the systemic vascular resistance index using a FloTrac(R) sensor. J Cardiothorac Vasc Anesth. 2013 Aug;27(4):696-702. doi: 10.1053/j.jvca.2012.11.019. Epub 2013 May 3. PMID 23648081
- [Background] Torella F, McCollum CN. Regional haemoglobin oxygen saturation during surgical haemorrhage. Minerva Med. 2004 Oct;95(5):461-7. PMID 15467521
- [Background] Uski T, Andersson KE, Brandt L, Edvinsson L, Ljunggren B. Responses of isolated feline and human cerebral arteries to prostacyclin and some of its metabolites. J Cereb Blood Flow Metab. 1983 Jun;3(2):238-45. doi: 10.1038/jcbfm.1983.32. PMID 6341384
- [Background] Wienecke T, Olesen J, Oturai PS, Ashina M. Prostacyclin (epoprostenol) induces headache in healthy subjects. Pain. 2008 Sep 30;139(1):106-116. doi: 10.1016/j.pain.2008.03.018. Epub 2008 May 2. PMID 18450380

RESULTS

PARTICIPANT FLOW:
Groups:
- Study of Cerebral Blood Flow: Patients undergoing oesophageal- or ventricular resection (n=30)
  Study of cerebral blood flow: Measurements are conducted from before induction of anaesthesia and until 2 hours after the start of surgery and include internal carotid artery blood flow, mean arterial pressure, heart rate, stroke volume, cardiac output, total peripheral resistance, forehead skin blood flow and haemoglobin concentrations, depth of anaesthesia, and frontal lobe, skin, and muscle oxygenation. Further measurements are conducted during hyperventilation before induction of anaesthesia and during hypo-, normo- and hypercapnia during anaesthesia.
  Blood samples are obtained from the arterial line for evaluation of the arterial CO2 tension and markers of mesenteric traction syndrome. Total volume of blood sampled is less than 75 ml.
Period: Overall Study
Arm/Group | Study of Cerebral Blood Flow
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 27
Internal carotid artery blood flow during anesthesia-induced hypotension [Mean (Standard Deviation); unit: ml/min] | 193 (41)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Internal Carotid Artery Blood Flow by Treatment of Anaesthesia-induced Hypotension
Description: Unilateral internal carotid artery blood flow [ml/min] assessed by duplex ultrasound.
Time Frame: Two measurements; one measurement during anaesthesia-induced hypotension (mean arterial pressure < 65 mmHg) before administration of phenylephrine and one measurement 3-5 min after administration of phenylephrine.
Measure: Mean (95% Confidence Interval); unit: ml/min
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 24
ml/min | 27 [3 to 51]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p = 0.0276, repeated measure mixed model

2. Secondary Outcome: Changes in Internal Carotid Artery Blood Flow by Induction of Anaesthesia.
Description: Unilateral internal carotid artery blood flow [ml/min] assessed by duplex ultrasound.
Time Frame: Two measurements; one measurement 5-10 min before induction of anaesthesia and one measurement 5-20 min after induction of anaesthesia.
Measure: Mean (95% Confidence Interval); unit: ml/min
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 30
ml/min | -144 [-168 to -121]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p < 0.0001, repeated measure mixed model

3. Secondary Outcome: Association by Multiple Regression Between Changes in Internal Carotid Artery Blood Flow, Mean Arterial Pressure and Cardiac Output by Treatment of Anaesthesia-induced Hypotension.
Description: Association by multiple regression between changes in unilateral internal carotid artery blood flow [ml/min] as outcome variable and changes in mean arterial pressure [mmHg] and cardiac output [l/min] as covariates.
  Internal carotid artery blood flow [ml/min] was assessed by duplex ultrasound. Mean arterial pressure [mmHg] was recorded by a transducer connected to an arterial line. Cardiac output [l/min] was evaluated by pulse contour analysis (Modelflow) that estimates cardiac output by analysis of the arterial pressure curve taking age, gender, height and weigth into account.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: ml/min
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 24
ml/min | 376 (724)
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p = 0.6025, Regression, Linear

4. Secondary Outcome: Changes in Frontal Lobe Oxygenation by Development of Mesenteric Traction Syndrome (MTS).
Description: Near-infrared spectroscopy determined frontal lobe oxygenation [%] as compared between those patients who develop a MTS (defined as flushing within 60 min after the start of surgery) and those who do not. An effect of a MTS was evaluated by a repeated measure mixed model with the fixed effects time point, group according to development of MTS, and interaction between time and group. The reported result is the interaction factor for the time point 0 min after flushing and 20 min after the start of surgery in patients who did not develop MTS.
Time Frame: Six measurements during anaesthesia; 5 min before and after incision and 0, 20, 40, and 70 min after flushing and 20, 40, 60, and 90 min after the start of surgery in those patients who do not develop mesenteric traction syndrome.
Measure: Mean (95% Confidence Interval); unit: oxygenation [%]
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
oxygenation [%] | 2 [-2 to 7]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p = 0.3213, repeated measure mixed model

5. Secondary Outcome: Changes in Forehead Skin Blood Flow by Development of Mesenteric Traction Syndrome (MTS).
Description: Forehead skin blood flow [PU] assessed by laser Doppler flowmetry as compared between those patients who develop mesenteric traction syndrome (defined as flushing within 60 min after the start of surgery) and those who do not. Laser Doppler flowmetry applies a laser placed on the forehead that penetrates the skin and is scattered with a Doppler shift by the red blood cells and return to a detector that evaluates the amount of backscattered light and Doppler shift. An effect of a MTS was evaluated by a repeated measure mixed model with the fixed effects time point, group according to development of MTS, and interaction between time and group. The reported result is the interaction factor for the time point 0 min after flushing and 20 min after the start of surgery in patients who did not develop MTS.
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: PU
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
PU | 126 [57 to 195]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p = 0.0005, repeated measure mixed model — The reported p-value was calculated

6. Secondary Outcome: Changes in Forehead Skin Oxygenation by Development of Mesenteric Traction Syndrome (MTS).
Description: Forehead skin oxygenation [%] assessed by laser Doppler flowmetry as compared between those patients who develop a MTS (defined as flushing within 60 min after the start of surgery) and those who do not. An effect of a MTS was evaluated by a repeated measure mixed model with the fixed effects time point, group according to development of MTS, and interaction between time and group. The reported result is the interaction factor for the time point 0 min after flushing and 20 min after the start of surgery in patients who did not develop MTS.
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: oxygenation [%]
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
oxygenation [%] | -2 [-9 to 5]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p = 0.5404, repeated measure mixed model

7. Secondary Outcome: Changes in Internal Carotid Artery Blood Flow by Development of Mesenteric Traction Syndrome (MTS).
Description: Unilateral internal carotid artery blood flow [ml/min] assessed by duplex ultrasound as compared between those patients who develop a MTS (defined as flushing within 60 min after the start of surgery) and those who do not. An effect of a MTS was evaluated by a repeated measure mixed model with the fixed effects time point, group according to development of MTS, and interaction between time and group. The reported result is the interaction factor for the time point 0 min after flushing and 20 min after the start of surgery in patients who did not develop MTS.
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ml/min
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
ml/min | -3 [-40 to 35]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p = 0.8947, repeated measure mixed model

8. Secondary Outcome: Changes in the CO2 Reactivity of the Internal Carotid Artery From Before to After Induction of Anaesthesia.
Description: Unilateral internal carotid artery blood flow [ml/min] assessed by duplex ultrasound and arterial CO2 tension (PaCO2) [kPa] was evaluated by gas analysis. Changes in PaCO2 are guided by evaluation of end-tidal CO2 tension.
  The CO2 reactivity to hypocapnia when awake and during anaesthesia is calculated as the percentage change in internal carotid artery blood flow per kPa change in PaCO2. The CO2 reactivity when awake and when anaesthetized is compared.
Time Frame: Four measurements; before induction of anaesthesia during normoventilation and during hyperventilation to reduce PaCO2 by 1.5 kPa and during anaesthesia at a PaCO2 at the value before induction of anaesthesia and 1.5 kPa below that value.
Population: Comparison of reactivity to hypocapnia when awake and during anaesthesia was evaluated by a linear mixed model with the relative change in ICA flow as outcome and fixed effects were the change in PaCO2 and an interaction factor for the difference between awake and anaesthesia. The reported result is the interaction factor.
Measure: Mean (95% Confidence Interval); unit: %/kPa
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
%/kPa | 7.4 [2.1 to 12.7]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p = 0.0068, Linear mixed models

9. Secondary Outcome: Changes in Heart Rate From Baseline Before Induction of Anaesthesia.
Description: Heart rate [bpm] as recorded continuously by a transducer connected to an arterial line.
Time Frame: Continuous measurements from before induction of anaesthesia and until 2 hours after start of surgery.
Measure: Mean (95% Confidence Interval); unit: beats/min
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
beats/min | -13 [-17 to -9]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p < 0.0001, repeated measure mixed model

10. Secondary Outcome: Changes in Mean Arterial Pressure From Baseline Before Induction of Anaesthesia.
Description: Mean arterial pressure [mmHg] as recorded continuously by a transducer connected to an arterial line.
Time Frame: Continuous measurements from before induction of anaesthesia and until 2 hours after start of surgery.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
mmHg | -41 [-47 to 35]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p < 0.0001, Mixed Models Analysis

11. Secondary Outcome: Changes in Cardiac Output From Baseline Before Induction of Anaesthesia.
Description: Cardiac output [l/min] as evaluated continuously by pulse contour analysis of the arterial pressure curve (Modelflow).
Time Frame: Continuous measurements from before induction of anaesthesia and until 2 hours after start of surgery.
Measure: Mean (95% Confidence Interval); unit: l/min
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
l/min | -2.7 [-3.4 to -2.0]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p < 0.0001, repeated measure mixed model

12. Secondary Outcome: Changes in Stroke Volume From Baseline Before Induction of Anaesthesia.
Description: Stroke volume [ml] as evaluated continuously by pulse contour analysis of the arterial pressure curve (Modelflow).
Time Frame: Continuous measurements from before induction of anaesthesia and until 2 hours after start of surgery.
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | Study of Cerebral Blood Flow
Number analyzed (Participants) | 27
ml | -24 [-34 to -14]
Statistical Analysis 1: Comparison: Study of Cerebral Blood Flow; Test type: Superiority; p < 0.0001, repeated measure mixed model

ADVERSE EVENTS:
Time Frame: Adverse event data were recorded during the patients stay in the operation room
Arm/Group | Study of Cerebral Blood Flow
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02951273/Prot_002.pdf
  • Statistical Analysis Plan (2017-11-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02951273/SAP_003.pdf